CLINICAL TRIAL: NCT05735158
Title: A Phase 2, Randomized, Placebo-controlled Study of Topical KB105, a Replication-defective, Non-integrating HSV-1 Vector Expressing Human Transglutaminase 1 (TGM1) for the Treatment of TGM1-deficient Autosomal Recessive Congenital Ichthyosis (ARCI)
Brief Title: Topical KB105 for the Treatment of TGM1-deficient Autosomal Recessive Congenital Ichthyosis (ARCI)
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Krystal Biotech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: KB105-02
Record Dates: First submitted 2023-02-09; First posted 2023-02-21 (Actual); Last update posted 2023-02-23 (Actual); Status verified 2023-02

CONDITIONS: Autosomal Recessive Ichthyosis

STUDY DESIGN:
Intervention Model Description: An intra-participant parallel study. Matched target areas will be randomized within the participant, such that one target area receives KB105 and the other target area will receive placebo. An additional target area may be selected to receive open-label treatment with KB105.
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- KB105 (Experimental): Weekly topical application
  Interventions: Biological: KB105
- Placebo (Placebo Comparator): Weekly topical application
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: KB105 — Replication-defective, non-integrating HSV-1 vector expressing TGM1 formulated as a topical gel
  Arms: KB105
Other: Placebo — Visually matched excipient gel
  Arms: Placebo

SUMMARY:
KB105-02 is an intrasubject randomized, placebo-controlled, double-blind study to evaluate the safety and efficacy of KB105 in children and adults with autosomal recessive congenital ichthyosis (ARCI).

ELIGIBILITY:
Key Inclusion Criteria:

1. Subject, or legally authorized representative, must be willing and able to give informed consent/assent
2. Aged ≥6 months
3. A genetically confirmed diagnosis of TGM1-deficient ARCI
4. Clinical diagnosis of lamellar ichthyosis
5. Two target areas located on similar anatomical regions with the same scaling severity by IGA and scaling severity ≥3
6. Subjects taking systemic retinoids must be on a stable regimen for at least 4 weeks and agree to continue to take the medication consistently throughout the study. If the subject prefers to withhold systemic retinoids during the study, then a minimum 4-week washout period is required
7. Clinically stable and in good general health

Key Exclusion Criteria:

1. Subject has a physical condition or other dermatological disorder (e.g., atopic, seborrheic, or contact dermatitis, psoriasis, tinea infections, etc.) which, in the Investigator's opinion, might impair evaluation of the target areas or which exposes the subject to unacceptable risk by study participation
2. Participation in another clinical study or treatment with an investigational agent within 30 days or 5 half-lives, whichever is longer
3. Any condition or illness (including a history or current evidence of substance abuse or dependence) that, in the opinion of the Investigator, would impact a subject's ability to complete all study-related procedures and/or poses an additional risk to the assessment of safety of KB105
4. Women who are pregnant or nursing
5. Subject who is unwilling to comply with contraception requirements per protocol
6. Subject is known to be noncompliant or is unlikely to comply with the requirements of the study protocol in the opinion of the Investigator

Min Age: 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2023-03 (Estimated); Primary Completion 2024-03 (Estimated); Study Completion 2024-04 (Estimated)

PRIMARY OUTCOMES:
Composite Investigator's Global Assessment (IGA) Responder (Comparison of proportion of responder KB105 target areas to responder placebo target areas) | Week 9
  Responder target areas are defined as:
  Target areas with ≥2 point reduction from baseline on IGA scaling severity at Week 9 or Target areas with ≥1 point reduction from baseline on IGA scaling severity for 2 consecutive weeks (Week 8 and Week 9)

SECONDARY OUTCOMES:
Composite regional Visual Index of Ichthyosis Severity (VIIS) responder (Comparison of proportion of responder KB105 target areas to responder placebo target areas) | Week 9
  Responder target areas are defined as:
  Target areas with ≥2 point reduction from baseline on VIIS scaling score at Week 9 or Target areas with ≥1 point reduction from baseline on VIIS scaling score for 2 consecutive weeks (Week 8 and Week 9)
Visual Index of Ichthyosis Severity score change from baseline | Up to 11 weeks
  Change from baseline in regional Visual Index of Ichthyosis Severity (VIIS) scaling scores, where 0 is normal and 4 is severe
Investigator's Global Assessment change from baseline | Up to 11 weeks
  Change from baseline in Investigator's Global Assessment (IGA) scaling severity scores, where 0 is clear and 4 is severe
Investigator's Global Assessment (IGA) 2 point responder | Week 9
  Comparison of proportion of KB105 and placebo target areas with ≥2 point reduction from baseline on IGA scaling severity at Week 9
Investigator's Global Assessment (IGA) 1 point responder | Week 9
  Comparison of proportion of KB105 and placebo target areas with ≥1 point reduction from baseline on IGA scaling severity for 2 consecutive weeks (Week 8 and Week 9)
Visual Index of Ichthyosis Severity (VIIS) 2 point responder | Week 9
  Comparison of proportion of KB105 and placebo target areas with ≥2 point reduction from baseline on regional VIIS scaling severity at Week 9
Visual Index of Ichthyosis Severity (VIIS) 2 point responder | Week 9
  Comparison of proportion of KB105 and placebo target areas with ≥1 point reduction from baseline on regional VIIS scaling severity for 2 consecutive weeks (Week 8 and Week 9)

CONTACTS AND LOCATIONS:
Locations (1):
- Mission Dermatology, Rancho Santa Margarita, California, United States